CLINICAL TRIAL: NCT05469321
Title: A Retrospective Study of Neurological Impairment in a Young Population Exposed to Recreational Nitrous Oxide
Brief Title: Neurological Impairment in a Young Population Exposed to Recreational Nitrous Oxide
Acronym: N2O
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: Local/2022/II-03
Record Dates: First submitted 2022-07-19; First posted 2022-07-21 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Neuropathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: patients presenting to the CHU of Nîmes for an acute or subacute neurological picture after having consumed N2O.
  Interventions: Other: None, pure observationnal study

INTERVENTIONS:
Other: None, pure observationnal study — None, pure observational study following the usual management of the patients

SUMMARY:
Nitrous oxide (N2O) is a colorless, flammable, analgesic gas used in surgery and dentistry. The consumption of N2O has increased among young French people aiming to relax because of its short-lived neuropsychological effect (euphoria, depersonalization, analgesia) and its wide availability on the market.

It can be responsible in case of prolonged use and overdose of a vitamin B12 deficiency with possible neuropsychiatric complications: sensitivomotor neuropathy, myelopathy, behavioral and cognitive disorders of acute or sub-acute installation.

N2O inhibits the activitý of methionine synthase, decreases the activitý of methylmalonyl-CoA mutase leading to vitamin B12 deficiency but in addition to the interference with vitamin B12 metabolism there seems to be a direct toxicity of N20.

Myelin alteration was the typical electromyography finding but new axonal profiles were also described. Since myelopathy affects both the posterior and lateral cords, combined spinal cord sclerosis is the most common location of injury associated with N2O intoxication.

ELIGIBILITY:
patients presenting to the CHU of Nîmes with an acute or sub-acute neurological picture after having consumed N2O

-

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients presenting to the CHU of Nîmes with an acute or sub-acute neurological picture after having consumed N2O
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-08-22 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
MRC score | baseline
  MRCss - Medical Research Council sum score : This score assigns a rating to each muscle group: "0" = absence of visible contraction visible contractions, " 1 " = visible contractions without movement of limbs, " 2 " = insufficient 2" = insufficient movements to overcome weightlessness, "3" = movements to overcome weightlessness, "4" = movements against weightlessness and resistance, "5" = normal muscle strength.
Romberg score | Baseline
  A positive Romberg test means the presence of sensory ataxia
INCAT Sensory Sum score (ISS) | Baseline
  grades from 0 (no involvement) to 20 (severe involvement)
ONLS - Overall Neuropathy Limitations Scale | Baseline
  Overall Neuropathy Limitation Scale = arm scale (range 0 to 5) + leg scale (range 0 to 7); (range: 0 (no disability) to 12 (maximum disability)
Rankin score | Baseline
  disability measurement score from 0 (none) to 6 (death)
vitamin B12 level | baseline
  vitamin B12 level in µmom/L
methyl malonic acid level | baseline
  methyl-malonic acid level
electroneuromyogram | baseline
  Normal Yes/No
Cerebral MRI | baseline
  lesions yes/No
Pan-medullary MRI | baseline
  lesions yes/No

CONTACTS AND LOCATIONS:
Overall Officials: Anissa MEGZARI, Study Director — Centre Hospitalier Universitaire de Nīmes
Locations (1):
- CHU de Nîmes, Nîmes, France